CLINICAL TRIAL: NCT06452251
Title: Vitamin-D Insufficiency Leads to Interleukin-10 Reduction in Peri-implant Tissues: A Case-Control Study
Brief Title: Vitamin-D Insufficiency and Implants
Status: Completed | Type: Observational
Sponsor: Vesile Elif Toy (Other)
Collaborators: Inonu University (Other)
Responsible Party: Sponsor-Investigator, Vesile Elif Toy, Assisstant professor, Inonu University
Organization: Inonu University (Other)
Other Study IDs: TSA-2022-2992
Record Dates: First submitted 2024-05-30; First posted 2024-06-11 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Vitamin D Deficiency; Osseointegration Failure of Dental Implant; Peri-Implantitis
Keywords: RANKL; calcium; IL-10; vitamin D; osseointegration
MeSH Terms: conditions — Vitamin D Deficiency; Peri-Implantitis | interventions — Radiography, Panoramic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- vitamin D sufficient: Vitamin D sufficient group (Group S) >20 ng/ml threshold was determined as sufficiency,
  Interventions: Diagnostic Test: OPG, OC, RANKL, IL-10, IL-1β, Ca, TNF-α and Caspase-1 ELISA; Diagnostic Test: Resonance Frequency Analysis; Diagnostic Test: Periodontal clinical examination; Procedure: Dental implant placement and bone sample collection; Procedure: Gingival Crevicular Fluid Sampling
- vitamin d insufficient: Vitamin D insufficient group (Group IN-S) 12-20 ng/mol was determined as insufficiency.
  Interventions: Diagnostic Test: OPG, OC, RANKL, IL-10, IL-1β, Ca, TNF-α and Caspase-1 ELISA; Diagnostic Test: Resonance Frequency Analysis; Diagnostic Test: Periodontal clinical examination; Procedure: Dental implant placement and bone sample collection; Procedure: Gingival Crevicular Fluid Sampling

INTERVENTIONS:
Diagnostic Test: OPG, OC, RANKL, IL-10, IL-1β, Ca, TNF-α and Caspase-1 ELISA — The levels of OPG, OC, RANKL, IL10, IL1β, Ca, TNF-α and Caspase1 in bone and PICF of patients with or without Vitamin D sufficiency were measured by ELISA.
Diagnostic Test: Resonance Frequency Analysis — Implant stability was measured by a device (Penguin RFA, Integration Diagnostics, Sweden) based on Resonance Frequency Analysis (RFA) and categorized by Implant Stability Quotient (ISQ) scale.
Diagnostic Test: Periodontal clinical examination — Clinical periodontal indices including plaque index (PI) (Silness and Löe 1964), gingival index (GI) (Löe 1967), probing depth (PD), and bleeding on probing (BOP) (Ainamo and Bay 1975) were recorded using a Williams periodontal probe. The BOP percentage (%) was calculated by dividing the number of bleeding sites by the total number of sites examined.
Procedure: Dental implant placement and bone sample collection — All patients were received by a single examiner a bone level implant (standard type and Sandblasted, Large-grit, Acid-etched surface) (Implant Swiss, Yverdon, Switzerland).
Procedure: Gingival Crevicular Fluid Sampling — One month after the healing caps were inserted, peri-implant crevicular fluid (PISF) samples were collected from 6 different sides of each implant. Before sampling, the area was isolated and dried, and paper strips were gently kept in periimplant sulcus for 30 seconds. Strips with blood or saliva contamination were discarded. PISF volumes of each strip were measured by a device (Periotron 8,010, Oraflow Inc, USA). Strips were then pooled, and inserted into tubes. PISF was recovered from paper strips through agitation in phosphate buffer saline (50 mM Tris-HCl, 5 mM CaCl2, 0.2 M NaCl,pH 7.5). All samples were stored at -80C until the day of analysis.

SUMMARY:
Vitamin D is important for bone health, immune function, and inflammation, along with dental implant success. The study aimed to assess bone markers and cytokine levels in patients with and without vitamin D insufficiency to better understand the effects of vitamin D levels on dental implant integration. The study included 42 patients in 2 groups; with insufficient (Group IN-S; n=21) and sufficient (Group S; n=21) levels of vitamin D. Bone remodelling, proinflammatory and antiinflammatory markers were analyzed in bone and peri-implant crevicular fluid (PICF) using enzyme-linked immunosorbent assay (ELISA) and results were reported as concentration and total amount.

DETAILED DESCRIPTION:
Background: Vitamin D is crucial for bone mineralization and plays a significant role in immune and inflammatory responses. Its deficiency is highly prevalent and might alter osseointegration of dental implants. Since successful osseointegration is a critical aspect of implant survival and the effects of vitamin D on implant osseointegration have not been well documented, the aim of this study was to evaluate bone markers and cytokine levels of patients with or without vitamin D insufficiency. Methods: A total of 42 patients were included and divided into two groups: Vitamin D insufficient (Group IN-S; n=21) and Vitamin D sufficient (Group S; n=21). Besides clinical periodontal parameters and implant stability measurements, bone and peri-implant crevicular fluid (PICF) levels of Receptor Activator of Nuclear Factor Kappa B Ligand (RANKL), osteoprotegerin (OPG), osteocalcin (OC), calcium (Ca), tumour necrosis factor alpha (TNF-α), Interleukin 1β (IL-1β), caspase-1 and Interleukin 10 (IL-10) were determined by enzyme-linked immunosorbent assay (ELISA). Results were represented as concentration and total amount.

ELIGIBILITY:
Inclusion Criteria:

Being volunteer to participate in the study, For the Vitamin D sufficient group (Group S) having a vitamin D level >20 ng/ml; and 12-20 ng/ml for Vitamin D insufficient group (Groups IN-S).

Having sufficient bone height and width at the edentulous areas, Not having a systemic disease that may adversely affect osseointegration, Not smoking Maintaining oral hygiene

Exclusion Criteria:

Vitamin D deficient patients (<12 ng/ml), already using vitamin D supplements Presence of any systemic disease, such as uncontrolled diabetes, that may affect implant success, Smoking, Presence of untreated periodontitis, Previous exposure to radiotherapy in the head and neck area, Presence of osteoporosis or other metabolic bone diseases, Usage of oral/intravenous bisphosphonates, History of bone grafting and/or sinus lift, Long-term corticosteroid usage.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: For the Vitamin D sufficient group (Group S) >20 ng/ml threshold was determined as vitamin D sufficient, and Vitamin D insufficient group (Groups IN-S) 12-20 ng/mol was determined as insufficient. Vitamin D deficient patients (<12 ng/ml), already using vitamin D supplements, were not included in the current study.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
change from baseline to 3 months for IL10 and RANKL | 0 to 3 months
  PICF and bone levels of markers were measured at baseline and at 3 months in both groups
change from baseline to 3 months for RFA | 0 to 3 months
  Measurement of primary and secondary implant stability were performed at baseline and at 3 months in both groups

CONTACTS AND LOCATIONS:
Overall Officials: Vesile E Toy, Phd, Principal Investigator — Inonu University
Locations (1):
- Inonu University, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Study data will be shared upon request by primary investigator Dr Vesile Elif toy elif.toy@inonu.edu.tr
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data is currently available.
Access Criteria: Individual participant data can be shared upon reasonable request.

REFERENCES:
- [Background] Akkaya HU, Yilmaz HE, Narin F, Saglam M. Evaluation of galectin-3, peptidylarginine deiminase-4, and tumor necrosis factor-alpha levels in gingival crevicular fluid for periodontal health, gingivitis, and Stage III Grade C periodontitis: A pilot study. J Periodontol. 2022 Jan;93(1):80-88. doi: 10.1002/JPER.21-0137. Epub 2021 May 10. PMID 33913157
- [Background] Kwiatek J, Jaron A, Trybek G. Impact of the 25-Hydroxycholecalciferol Concentration and Vitamin D Deficiency Treatment on Changes in the Bone Level at the Implant Site during the Process of Osseointegration: A Prospective, Randomized, Controlled Clinical Trial. J Clin Med. 2021 Feb 2;10(3):526. doi: 10.3390/jcm10030526. PMID 33540512
- [Background] Franco-Topete R, Zepeda-Nuno JS, Zamora-Perez AL, Fuentes-Lerma MG, Gomez-Meda BC, Guerrero-Velazquez C. IFN-gammaR2 is strongly expressed on endothelial cells of gingival tissues from patients with chronic periodontitis. J Appl Oral Sci. 2018 Oct 4;26:e20170291. doi: 10.1590/1678-7757-2017-0291. PMID 30304122